CLINICAL TRIAL: NCT02742753
Title: Impact of Pneumococcal Conjugate Vaccines on Otitis Media and Acute Otitis Media in Swedish Children
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 203129
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Acute Otitis Media; Otitis Media
Keywords: Otitis; Vaccine; Sweden; Database
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Study cohort: The Total population will include all subjects included in the study. Only aggregated information will be collected for these subjects.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data will be collected retrospectively linking regional patient-level data prospectively captured in real-world clinical setting with mandatory national healthcare registries from 2004 to 2013.

SUMMARY:
The goal of this study is to look at the effect of pneumococcal conjugate vaccines (PCV) on physician-diagnosed otitis media (OM) and acute otitis media (AOM) incidence in Swedish children by collecting and analyzing patient level observational data already available in existing regional and national databases.

ELIGIBILITY:
Inclusion Criteria:

Data from all children ≤ 5 years old in VGR and Skåne in each year during the study period (2004 - 2013)

Exclusion Criteria:

Not Applicable

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children living in the county councils of VGR and Skåne during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the impact of PCVs by describing, separately for Skåne and VGR (Västra Götalandsregionen), trends over time in the incidence of OM and AOM among children during the pre-PCV, PCV7, and Synflorix®/PCV13-eras | During 10 years: from January 1, 2004 to December 31, 2013
  A step-wise approach will be applied: 1. Descriptive analyses to assess any trends in OM and AOM incidence, any seasonality (repeating pattern of incidence related to time such as seasons, quarters and months), the order of seasonality, extreme observations/outliers, whether incidence trends include abrupt changes. 2. If trends or seasonality are identified, a time series analysis will be conducted in 2 steps. a. Time series analysis of monthly incidence, using smoothing technique to estimate differences in pre-PCV, PCV7, and Synflorix®/PCV13 vaccination periods. b. Interrupted time-series analysis if the above steps show any differences in pre- and post- vaccination introduction periods. Diagnoses of AOM recorded under the ICD-10 code H66 (suppurative and unspecified OM) and ICD-10 H66.0 (acute suppurative OM); Chronic OM under ICD-10 code H66.3 (other chronic suppurative OM) and other OM underICD-10 code H66.9 (OM unspecified) and H65 (non-suppurative OM).

SECONDARY OUTCOMES:
Assessment of the impact of PCVs by describing trends over time in the rate of antibiotics dispensed for OM and AOM diagnoses among children with OM or AOM | During 10 years: from January 1, 2004 to December 31, 2013
  The impact of PCV will be investigated by looking at trends over time in the rate of antibiotics* dispensed due to an OM or AOM diagnosis for the two counties separately. The analysis of rate of antibiotic use will be performed in two steps as: Descriptive statistics for the number of dispensed antibiotics. Time series analysis for the incidence of dispensed antibiotics. *Date of an antibiotic dispensed within 7 days of a registered diagnosis code (ICD-10 code H65, H66, H66.0, H66.3, H66.9).
Assessment of the the impact of PCVs by describing trends over time in the rate of tympanostomy tube insertions among children with OM and AOM | During 10 years: from January 1, 2004 to December 31, 2013
  The rate of tympanostomy tube insertions* among children with OM or AOM will also be analyzed in the same way as the analysis of frequency of antibiotics dispensed. *Date of Tympanostomy tube placement procedure (KVA DCD10).
Assessment of the impact of PCVs by describing the trends over time in the incidence of severe AOM (Medical Products Agency 2010, Lieberthal 2013) among children | During 10 years: from January 1, 2004 to December 31, 2013
  The impact of PCVs on the incidence of severe AOM among children will be analysed with a step-wise time series analysis approach, which is described for the primary outcome. Severe AOM defined as: -Children diagnosed with AOM with presence of moderate to severe otalgia or fever ≥ 39° C, or -Children with ≥3 diagnoses of AOM in a 6-month period or ≥4 AOM diagnoses in a 12-month period, or-Children reported with hospitalization due to AOM or any documented evidence of IV infusion of antibiotics in hospital.
Assessment of the Costs for OM and AOM-related healthcare resource utilization | During 10 years: from January 1, 2004 to December 31, 2013
  Cost dispersion statistics (mean, median, standard deviation, minimum, maximum, variance) will be calculated. Direct costs for OM and AOM will be calculated by including healthcare resource utilization for each child as the count of antibiotic prescriptions filled for OM and AOM, and use of medical services, such as visits to the general practitioner, visits to the hospital, procedure costs (tympanostomy tube placements, myringotomies and IV antibiotics administrations) and length of hospital stay during the follow-up period. Cost for all health care visits and procedures will be calculated using the number of registered events multiplied by a unit cost based on public price lists for that particular visit or procedure.
Assessment of possible individual-level predictors for the time to the first OM or AOM diagnosis | During 10 years: from January 1, 2004 to December 31, 2013
  The following analysis will be conducted to understand individual-level factors that impacts OM and AOM rates and time to first incidence of an OM or an AOM separately for each county council. A survival analysis will be conducted to assess predictors of the time to first OM or AOM using a left censored Cox proportional hazards model.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edmondson-Jones M, Dibbern T, Hultberg M, Anell B, Medin E, Feng Y, Talarico C. The effect of pneumococcal conjugate vaccines on otitis media from 2005 to 2013 in children aged </=5 years: a retrospective cohort study in two Swedish regions. Hum Vaccin Immunother. 2021 Feb 1;17(2):517-526. doi: 10.1080/21645515.2020.1775455. Epub 2020 Jun 23. PMID 32574101
- See also: Results for study 203129 can be found on the GSK Clinical Study Register — https://www.gsk-studyregister.com/study/5586